CLINICAL TRIAL: NCT06198920
Title: Atherosclerotic Pathology of the Superficial Femoral Arteries: Study and Patient-specific Prediction of the Fatigue Behavior of Peripheral STENt in Nitinol Via Mathematical Modeling. Prospective Enrollment
Brief Title: Fatigue Behavior of Peripheral STENt of the Superficial Femoral Artery
Acronym: FASTEN-PRO
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Daniela Mazzaccaro, Vascular Surgeon, Researcher, PI, IRCCS Policlinico S. Donato
Other Study IDs: FASTEN-PRO V1 - 78/int/2017
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Atherosclerosis; Stent Complication
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Stenting of the superficial femoral artery — Submitted to stenting of the superficial femoral artery for stenosis or occlusion causing intermittent claudication or critical limb ischemia

SUMMARY:
Endovascular treatment of superficial femoral artery stenosis/obstruction is still the subject of debate in the scientific literature.

Previous clinical studies have in fact reported conflicting data regarding the benefits of implanting self-expanding Nitinol stents in the superficial femoral artery district compared to simple percutaneous transluminal angioplasty. Invariably, patient comorbidities and anatomic characteristics of the lesions appear to be important factors influencing procedural success and one-year patency rates. Additionally, there are concerns regarding the potential clinical impact of stent fractures, reported at rates ranging from 12% to 37.2% at one year.

Despite the improved outcomes seen with newer Nitinol stent designs, the primary limitations of stenting in the superficial femoral artery are the use of multiple overlapping stents or long stents and the associated potential rate of stent fracture resulting reocclusion of the treated superficial femoral artery and clinical worsening of patients who in most cases are initially treated for disabling claudication.

Being able to preoperatively determine in which patients there are risk factors prognostically associated with a higher rate of fracture/reocclusion could represent a help for the operator in choosing the best therapeutic strategy.

DETAILED DESCRIPTION:
The study involves the prospective collection of the following data:

* Preoperative: vessel diameters, plaque length, plaque type, percentage of stenosis, position of the stenosis. These data will be collected from the analysis of CT images, magnetic resonance imaging, color Doppler ultrasound or angiographies performed by patients in the diagnostic phase;
* Intraoperative: number and model (brand and size) of stent implanted, position of the stent. The stents used are those foreseen by the usual clinical practice of each center. In particular, the behavior of the following stents will be analysed:

or Absolute Pro® Vascular Self-Expanding Stent System - ABBOTT VASCULAR or S.M.A.R.T.® Flex Vascular Self-Expanding Stent - CORDIS or LifeStent® - BARD PV or Zilver® - COOK MEDICAL

- Follow-up: restenosis event, stent fracture event. In particular, the restenosis event will be defined by the presence of a reduction in the caliber of the vessel morphologically greater than 30% or with PVR (Peak Velocity Ratio = peak systolic velocity in correspondence with the stenosis/peak systolic velocity upstream in a non-stenotic tract ) recorded on color Doppler ultrasound > 2.4. The stent fracture event will be defined by the presence of discontinuity images in the stent structure itself. These data will be collected from the analysis of arterial color-Doppler ultrasound images of the lower limbs (reference investigation foreseen by the study) or other investigations (CT, magnetic resonance imaging, angiographies) performed by patients in the follow-up phase.

The mathematical model:

The computational analysis involves a reproduction via 3D model of the morphology of the pathological superficial femoral artery specific to the diagnostic data of the patients and the peripheral Nitinol stents used.

The recanalization/dilation and stenting treatment is simulated using a finite element model, taking into account the phases of the clinical procedure and the consequent cyclic stress conditions to which the device is subjected in vivo.

The results of the computational model are analyzed in order to obtain the state of stress acting on the device and evaluate its risk of breakage.

In particular, the models created to reproduce the cases of the study will be developed using a commercial software in which the collected pre- and intraoperative parameters are entered, and from which the prediction values of whether or not the superficial femoral stent will break will be extracted.

The prediction given by the mathematical model will be compared with the data actually observed during the 3-year follow-up.

The collected data will then be entered into a database and analyzed using the JMP 5.1.2 statistical software (S.A.S. Institute).

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 18 years) hospitalized in the Operating Units participating in the study and subjected to a recanalization/dilation and stenting procedure of the superficial femoral artery due to stenosis or obstruction of the same conditioning disabling claudication or critical ischemia of the lower limb (class 3-4-5-6 according to Rutherford).

Exclusion Criteria:

* minor patients (age <18 years);
* patients who have not given their consent to participate in the study;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by disabling intermittens claudication or critical limb ischemia due to stenosis/occlusion of the superficial femoral artery and treated with stenting of the superficial femoral artery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of Stenting failure (restenosis/occlusion/fracture) | 1 month
  determine the predictive capacity of a mathematical model developed by the LaBS (Laboratory of Biological Structure Mechanics), Department of Chemistry, Materials and Chemical Engineering "Giulio Natta", of the Polytechnic of Milan to predict the fracture of a stent positioned in superficial femoral artery for the treatment of stenosis/obstruction of the same in adult patients suffering from obliterating arterial disease of the lower limbs.
Rate of Stenting failure (restenosis/occlusion/fracture) | 6 months
  determine the predictive capacity of a mathematical model developed by the LaBS (Laboratory of Biological Structure Mechanics), Department of Chemistry, Materials and Chemical Engineering "Giulio Natta", of the Polytechnic of Milan to predict the fracture of a stent positioned in superficial femoral artery for the treatment of stenosis/obstruction of the same in adult patients suffering from obliterating arterial disease of the lower limbs.
Rate of Stenting failure (restenosis/occlusion/fracture) | 12 months
  determine the predictive capacity of a mathematical model developed by the LaBS (Laboratory of Biological Structure Mechanics), Department of Chemistry, Materials and Chemical Engineering "Giulio Natta", of the Polytechnic of Milan to predict the fracture of a stent positioned in superficial femoral artery for the treatment of stenosis/obstruction of the same in adult patients suffering from obliterating arterial disease of the lower limbs.
Rate of Stenting failure (restenosis/occlusion/fracture) | 24 months
  determine the predictive capacity of a mathematical model developed by the LaBS (Laboratory of Biological Structure Mechanics), Department of Chemistry, Materials and Chemical Engineering "Giulio Natta", of the Polytechnic of Milan to predict the fracture of a stent positioned in superficial femoral artery for the treatment of stenosis/obstruction of the same in adult patients suffering from obliterating arterial disease of the lower limbs.
Rate of Stenting failure (restenosis/occlusion/fracture) | 36 months
  determine the predictive capacity of a mathematical model developed by the LaBS (Laboratory of Biological Structure Mechanics), Department of Chemistry, Materials and Chemical Engineering "Giulio Natta", of the Polytechnic of Milan to predict the fracture of a stent positioned in superficial femoral artery for the treatment of stenosis/obstruction of the same in adult patients suffering from obliterating arterial disease of the lower limbs.

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Laird JR, Katzen BT, Scheinert D, Lammer J, Carpenter J, Buchbinder M, Dave R, Ansel G, Lansky A, Cristea E, Collins TJ, Goldstein J, Jaff MR; RESILIENT Investigators. Nitinol stent implantation versus balloon angioplasty for lesions in the superficial femoral artery and proximal popliteal artery: twelve-month results from the RESILIENT randomized trial. Circ Cardiovasc Interv. 2010 Jun 1;3(3):267-76. doi: 10.1161/CIRCINTERVENTIONS.109.903468. Epub 2010 May 18. PMID 20484101
- [Result] Chowdhury MM, McLain AD, Twine CP. Angioplasty versus bare metal stenting for superficial femoral artery lesions. Cochrane Database Syst Rev. 2014 Jun 24;2014(6):CD006767. doi: 10.1002/14651858.CD006767.pub3. PMID 24959692
- [Result] Soga Y, Iida O, Hirano K, Yokoi H, Nanto S, Nobuyoshi M. Mid-term clinical outcome and predictors of vessel patency after femoropopliteal stenting with self-expandable nitinol stent. J Vasc Surg. 2010 Sep;52(3):608-15. doi: 10.1016/j.jvs.2010.03.050. Epub 2010 Jun 22. PMID 20573476
- [Result] Krankenberg H, Schluter M, Steinkamp HJ, Burgelin K, Scheinert D, Schulte KL, Minar E, Peeters P, Bosiers M, Tepe G, Reimers B, Mahler F, Tubler T, Zeller T. Nitinol stent implantation versus percutaneous transluminal angioplasty in superficial femoral artery lesions up to 10 cm in length: the femoral artery stenting trial (FAST). Circulation. 2007 Jul 17;116(3):285-92. doi: 10.1161/CIRCULATIONAHA.107.689141. Epub 2007 Jun 25. PMID 17592075
- [Result] Scheinert D, Scheinert S, Sax J, Piorkowski C, Braunlich S, Ulrich M, Biamino G, Schmidt A. Prevalence and clinical impact of stent fractures after femoropopliteal stenting. J Am Coll Cardiol. 2005 Jan 18;45(2):312-5. doi: 10.1016/j.jacc.2004.11.026. PMID 15653033
- [Result] Schlager O, Dick P, Sabeti S, Amighi J, Mlekusch W, Minar E, Schillinger M. Long-segment SFA stenting--the dark sides: in-stent restenosis, clinical deterioration, and stent fractures. J Endovasc Ther. 2005 Dec;12(6):676-84. doi: 10.1583/05-1672.1. PMID 16363897
- [Result] Ihnat DM, Duong ST, Taylor ZC, Leon LR, Mills JL Sr, Goshima KR, Echeverri JA, Arslan B. Contemporary outcomes after superficial femoral artery angioplasty and stenting: the influence of TASC classification and runoff score. J Vasc Surg. 2008 May;47(5):967-74. doi: 10.1016/j.jvs.2007.12.050. Epub 2008 Apr 18. PMID 18372147
- [Result] Stabile E, Virga V, Salemme L, Cioppa A, Ambrosini V, Sorropago G, Tesorio T, Cota L, Popusoi G, Pucciarelli A, Biamino G, Rubino P. Drug-eluting balloon for treatment of superficial femoral artery in-stent restenosis. J Am Coll Cardiol. 2012 Oct 30;60(18):1739-42. doi: 10.1016/j.jacc.2012.07.033. Epub 2012 Oct 3. PMID 23040582
- [Result] Dordoni E, Meoli A, Wu W, Dubini G, Migliavacca F, Pennati G, Petrini L. Fatigue behaviour of Nitinol peripheral stents: the role of plaque shape studied with computational structural analyses. Med Eng Phys. 2014 Jul;36(7):842-9. doi: 10.1016/j.medengphy.2014.03.006. Epub 2014 Apr 12. PMID 24721457